CLINICAL TRIAL: NCT02748356
Title: The Impact of Self-Management With Probiotics on Urinary Symptoms and the Urine Microbiome in Individuals With Spinal Cord Injury (SCI) and Spina Bifida (SB)
Brief Title: Impact of Probiotics on Urinary Symptoms in Spinal Cord Injury SCI and SB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Children's National Research Institute (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5753
Record Dates: First submitted 2016-01-29; First posted 2016-04-22 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Spina Bifida; Spinal Cord Injury
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Spinal Dysraphism; Spinal Cord Injuries | interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individuals with Spina Bifida (Experimental): Lactobacillus rhamnosus GG
  Interventions: Drug: Lactobacillus

INTERVENTIONS:
Drug: Lactobacillus — Eligible patients will undergo 1 Lactobacillus pediatric dose (Culturelle GG 10 Billion live organisms) instillation by study personnel at the study site. For the intravesicular Lactobacillus instillation, the contents of 1 Lactobacillus capsule will be mixed into sterile 0.9% saline using an age-based estimate of bladder capacity. Similar to adults, this bladder instillation will represent 10% of the estimated maximum bladder volume based on age.
  Other Names: Culturelle

SUMMARY:
As a collaborative effort between MedStar National Rehabilitation Hospital (NRH), Children's National Medical Center (CNMC) Department of Urology, Children's Research Institute (CRI) Center for Genetic Medicine Research, Georgetown University, and MedStar Georgetown University Hospital, the overall objective of this study is to develop, validate, and assess a patient-initiated, probiotic-based, selfmanagement protocol that is initiated at the time of urinary symptoms. The self-management protocol will allow patients to manage urinary symptoms and avoid potentially unnecessary antibiotic use, and provide a readily-available means of maintaining health, function, and independence throughout the lifespan.

DETAILED DESCRIPTION:
Lower urinary symptoms are a common issue for individuals with neurogenic bladder, commonly occurring in the Spina bifida and Spinal Cord Injury population. In this study, probiotics will be introduced into the bladder to prevent UTIs. Introduction of probiotics will be determined by a validated symptom questionnaire (USQ-NB) and protocol (SMP-PRO).

This study will estimate the strength of the associations between successful implementation of the probiotic self-management program (USQ-NB and SMP-PRO) and urinary symptoms, bladder inflammation, and the urine microbiome. Investigators will conduct an 18-month study in which each participant will serve as his/her own control through 3 phases of study: 6-months usual care (baseline), 6-months probiotic intervention, and 6-months follow-up.

Participants will complete the Urinary Symptom Questionnaire weekly. After 6 months of baseline data collection, participants will receive the Lactobacillus (Culturelle GG, 20 billion live organisms for adults and 10 billion live organisms for children <18 years of age), will be instructed on preparation and intravesicular instillation of the Lactobacillus, and will have a tutorial with a fellow consumer on use of the patient-initiated protocol. The protocol and Lactobacillus bladder instillation instructions (including a step-by-step video) will be available on the study website for 24/7 access and written instructions will be provided at the time of instruction.

For the intravesicular Lactobacillus instillation, participants will be instructed to mix the contents into sterile saline. After mixing, participants will draw up the liquid Lactobacillus mixture into a 60cc catheter tip syringe and instill via the intermittent catheter after fully emptying the bladder. The amount instilled is determined by the age of the child. Participants will be instructed not to catheterize for at least 4 hours after the bladder instillation. Participants will receive 10 Culturelle GG at the beginning of the treatment phase. At the end of each month, the coordinator or RA will ask how many remaining tablets the participant has, and if needed dispense the next supply of 10 tablets. Participants will be instructed to complete the USQ-NB weekly.

If/when urinary symptoms occur, subjects will be instructed to follow the protocol to determine whether to initiate intravesicular Lactobacillus instillation or be evaluated by a physician. The self-management protocol will also direct them to discontinue Lactobacillus instillation or be evaluated by a physician if symptoms remit, persist (after 2 instillations), or worsen. The maximum number of instillations is 2 over 28 hours. If participants are directed by the self-management protocol to seek medical attention or s/he feels the need for medical evaluation, s/he will be advised to obtain care as they typically would by their health care provider. Participants will be supplied with letters to be brought to their health care provider notifying them of the study and requesting sharing of urinalysis and urine culture results with the research team. A verified UTI will include those that resulted in antibiotic treatment by a health care professional. An additional urine sample for metagenomics will either be left with the health care provider for pick up by the research team, brought to the research site, or obtained by the RA at a mutually convenient site.

After completion of the 6-month patient-initiated self-management protocol intervention period, participants will monitor symptoms weekly using the USQ-NB.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥6 years, and
2. Spina bifida and neuropathic bladder, as determined by the attending physician, and
3. Utilization of intermittent catheterization for bladder management, and
4. History of 2 or more urinary tract infections (UTIs) in the past year, and
5. Community dwelling.

Exclusion Criteria:

1. Has a known genitourinary pathology beyond neuropathic bladder (e.g. vesicoureteral reflux, bladder stones, kidney stones, etc), and/or
2. Uses prophylactic antibiotics, and/or
3. Uses intravesicular agents to reduce UTI (e.g. gentamycin), and/or
4. Has psychologic or psychiatric conditions influencing the ability to follow instructions, and/or
5. Participates in another study in which results would be confounded, and/or
6. Is pregnant or breastfeeding, and/or
7. Has a history of acquired or genetic immunodeficiencies, or active, acute or chronic serious infections (e.g. viral hepatitides, HIV/AIDs), and/or
8. Has cancer or an autoimmune disorder, and/or
9. Has a serious allergy to any component or excipients in the live bacterial combination product, and/or
10. Has had a change in neurologic status in the previous 2 weeks, and/or
11. Has taken antibiotic for any reason in the previous 2 weeks, and/or
12. Has a history of sensitivity or allergy to ampicillin or tetracycline, and/or
13. Has a current urinary tract infection or urinary tract infection within the previous 2 weeks (as defined by Infectious Diseases Society of America CAUTI Guidelines, 2010).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Pohl, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Individuals With Spina Bifida or Spinal Cord Injury: Lactobacillus instillation During intervention phase participants were instructed to instill a Lactobacillus solution via their intermittent catheter when they experienced cloudier or more bad- smelling, stronger, fouler or more pungent than their normal urine. These symptoms had to be experienced in the absence of fever, shaking chills, feeling unclear, foggy or confused, overall sense of discomfort, feeling more tired than usual, side pain in the lower back, tenderness to touch in the side of the low back, blood in urine, abdominal pain below, belly button, increase in muscle tightness or tone, autonomic dysreflexia, sense of unease.
Period: Overall Study
Arm/Group | Individuals With Spina Bifida or Spinal Cord Injury
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 6 children with Spina Bifida, 1 child SCI
Arm/Group | Individuals With Spina Bifida or Spinal Cord Injury
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Lactobacillus Safety
Description: Total Adverse Events (AE + Serious AE) per participants
Time Frame: months 1-18 of study
Measure: Mean (Standard Deviation); unit: Adverse Events
Arm/Group | Individuals With Spina Bifida or Spinal Cord Injury
Number analyzed (Participants) | 7
Adverse Events | .286 (.488)
Statistical Analysis 1: Comparison: Individuals With Spina Bifida or Spinal Cord Injury; Test type: Other — 1 sample t-test; p = 0.351, t-test, 2 sided; This is a single group comparison

2. Secondary Outcome: Lactobacillus Tolerability
Description: This is a one-item satisfaction rating. "While thinking only about the preceding 6-month time period: "can you estimate, using a scale from 0 to 100%, whether or not you would seek out this intervention and pay for it yourself if insurance did not pay for it?" Participants indicated their answer by moving a "slider" with three anchors: 0%=Would absolutely never do this; 50%=Might do this; 100%= Would absolutely do this. If a participant is less satisfied, their rating will be lower, and if they are more satisfied, the rating would be higher, but the item did not have options for "better" or "worse". This is not a published scale, we included this item in our general data collection.
  Ratings averaged over final 12 months of study (Satisfaction question was answered by study participants at 3 time points; 6 months, 12 months and 18 months)
Time Frame: months 7-18
Population: 5 out of 7 children instilled Lactobacillus at least once
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individuals With Spina Bifida or Spinal Cord Injury
Number analyzed (Participants) | 5
units on a scale | 73.6 (28.3)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the study (18 months)
Arm/Group | Individuals With Spina Bifida or Spinal Cord Injury
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individuals With Spina Bifida or Spinal Cord Injury (N=7)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Tethered spinal cord surgery (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02748356/Prot_SAP_000.pdf